CLINICAL TRIAL: NCT00938405
Title: Efficacy of Colesevelam in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Satish K. Garg, Professor of Medicine & Pediatrics, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSI-WCH-100
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 1; Hyperlipidemias
Keywords: type 1 diabetes mellitus; colesevelam; LDL; cholesterol; A1c; target range glucose values
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperlipidemias | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colesevelam HCl (Experimental): Beginning at Visit 1, two weeks after screening, subjects in the active treatment group will take 3.75 gms/day of colesevelam HCl in the form of three 625 mg tablets with lunch and dinner or six 625mg tablets once daily with dinner.
  Interventions: Drug: Colesevelam HCl
- Comparison group (Placebo Comparator): Beginning at Visit 1, two weeks after screening, subjects in the comparison group will be administered placebo, taking 3.75 gms/day of colesevelam HCl in the form of three 625 mg tablets with lunch and dinner or six 625mg tablets once daily with dinner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colesevelam HCl — 3.75 gms/day of colesevelam HCl in the form of three 625 mg tablets with lunch and dinner or six 625mg tablets once daily with dinner.
  Other Names: WELCHOL (colesevelam hydrochloride); Initial U.S. Approval: 2000
  Arms: Colesevelam HCl
Drug: Placebo — Placebo: 3.75 gms/day in the form of three 625 mg tablets with lunch and dinner or six 625mg tablets once daily with dinner.
  Arms: Comparison group

SUMMARY:
This is a prospective, randomized, double blind, parallel, placebo controlled clinical trial evaluating the efficacy of colesevelam HCl in reducing LDL in subjects with type 1 diabetes mellitus over a 12 week treatment period. The aim is to highlight the effect of colesevelam on LDL cholesterol and glycemia in a type 1 diabetic population. The colesevelam group is anticipated to demonstrate a mean reduction in LDL by 10% compared to the placebo group, indicated by A1c and glycemic target range CGM readings.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, parallel, placebo controlled clinical trial evaluating the efficacy of colesevelam HCl in reducing LDL in subjects with type 1 diabetes mellitus over a 12 week treatment period. Colesevelam is an orally administered bile acid sequestrant approved as an adjunct for diet and exercise for lowering incidence of hyperlipidemia, an important risk factor for long term cardiovascular health in the general population and people living with diabetes. Use of colesevelam has been shown to concurrently decrease low density lipoprotein cholesterol (LDL-C) and A1c in patients with type 2 diabetes. The exact mechanism is unknown. Our research aims to highlight the effect of colesevelam on LDL and glycemia in a type 1 diabetic population.

This single-center study will enroll a maximum of 40 patients with LDL-C > 100 and A1c values between 6.5-9%, who will be randomized in a 1:1 fashion to either the study drug or placebo. Visits will be conducted at screening, baseline, one month, two months, and three months. At home, subjects will take 3.75 gms/day of colesevelam HCl or placebo throughout the study duration. Laboratory analysis will be performed at various timepoints assessing A1c, fasting lipid panel, c-peptide, glucagon-like-peptide-1 (GLP-1), and glucose-dependent insulinotropic peptide (GIP). Continuous glucose monitoring (CGM) measurements will be obtained on all patients for one week before each monthly visit to assess for above target range (ATR), within target range (WTR), and below target range (BTR) glucose values and time spent in hyperglycemic and hypoglycemic excursions.

The colesevelam group is anticipated to demonstrate a mean reduction in LDL by 10% compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be on stable doses of insulin using MDI or CSII (Basal insulin- Lantus or Levemir; Bolus- Humalog, Novolog, Apidra, Humulin Regular), for three months prior to enrollment.
* Type 1 diabetes duration > 3 years.
* 6.5% ≤ A1c ≤ 9.0%.
* Male or female ≥ 18 and ≤ 65 years of age.
* Ability and willingness to adhere to the protocol including multiple daily oral doses of study drug or placebo and week-long CGM wear.
* LDL-C > 100 mg/dl.
* Willing to adhere to colesevelam dosage instructions, including administration of drugs with a known interaction at least 4 hours prior to colesevelam. Females using oral contraceptives containing ethinyl estradiol and norethindrone must be willing to administer their doses at least four hours prior to using colesevelam.

Exclusion Criteria:

* Advanced retinopathy needing laser procedure or vitrectomy.
* Unstable nephropathy (serum creatinine > 2.0 mg/dl or macroproteinuria (albumin excretion rate > 200 ug/ min).
* Any unexplained severe hypoglycemia within the last six months.
* BMI > 35.0.
* Currently on a pre-existing bile acid sequestrant therapy, glyburide, levothyroxine, phenytoin, or warfarin.
* Pregnant, planning a pregnancy, or not using an adequate method of birth control.
* Any other condition, as determined by the investigator, which could make the subject unsuitable for the trial, impairs the subject's suitability for the trial, or impairs the validity of the informed consent.
* Use of any medication known to modify glucose values other than insulin (i.e. corticosteroids or oral antidiabetics).
* A history of bowel obstruction.
* Serum triglyceride (TG) concentrations >500 mg/dL.
* A history of hypertriglyceridemia induced pancreatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate a 10% LDL reduction in type 1 diabetic subjects with initial LDL > 100 after twelve weeks in the colesevelam group. | 12 weeks of treatment

SECONDARY OUTCOMES:
To evaluate colesevelam use for glucose control as measured by A1c using a 0.4% confidence interval at baseline and after one, two, and three months of therapy. | 12 weeks of treatment.
To evaluate colesevelam use for non-inferiority of percent of target range glucose values and time spent in hyper- and hypoglycemic ranges as determined by CGM readings at baseline and after one, two, and three months of therapy. | 12 weeks of treatment.
In addition change in insulin dose at one, two and three months from baseline will be evaluated. | 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Satish K Garg, MD, Principal Investigator — University of Colorado Denver/ Barbara Davis Center for Diabetes
Locations (1):
- Barbara Davis Center for Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Background] Bays HE, Goldberg RB, Truitt KE, Jones MR. Colesevelam hydrochloride therapy in patients with type 2 diabetes mellitus treated with metformin: glucose and lipid effects. Arch Intern Med. 2008 Oct 13;168(18):1975-83. doi: 10.1001/archinte.168.18.1975. PMID 18852398
- [Background] Goldberg RB, Fonseca VA, Truitt KE, Jones MR. Efficacy and safety of colesevelam in patients with type 2 diabetes mellitus and inadequate glycemic control receiving insulin-based therapy. Arch Intern Med. 2008 Jul 28;168(14):1531-40. doi: 10.1001/archinte.168.14.1531. PMID 18663165
- [Background] Fonseca VA, Rosenstock J, Wang AC, Truitt KE, Jones MR. Colesevelam HCl improves glycemic control and reduces LDL cholesterol in patients with inadequately controlled type 2 diabetes on sulfonylurea-based therapy. Diabetes Care. 2008 Aug;31(8):1479-84. doi: 10.2337/dc08-0283. Epub 2008 May 5. PMID 18458145
- [Background] Goldfine AB, Fonseca VA. The use of colesevelam HCl in patients with type 2 diabetes mellitus: combining glucose- and lipid-lowering effects. Postgrad Med. 2009 May;121(3 Suppl 1):13-8. doi: 10.3810/pgm.2009.05.suppl53.288. PMID 19494473
- [Background] Staels B. A review of bile acid sequestrants: potential mechanism(s) for glucose-lowering effects in type 2 diabetes mellitus. Postgrad Med. 2009 May;121(3 Suppl 1):25-30. doi: 10.3810/pgm.2009.05.suppl53.290. PMID 19494475
- [Background] Garg SK, Kelly WC, Voelmle MK, Ritchie PJ, Gottlieb PA, McFann KK, Ellis SL. Continuous home monitoring of glucose: improved glycemic control with real-life use of continuous glucose sensors in adult subjects with type 1 diabetes. Diabetes Care. 2007 Dec;30(12):3023-5. doi: 10.2337/dc07-1436. Epub 2007 Sep 11. No abstract available. PMID 17848608